CLINICAL TRIAL: NCT01320943
Title: FINITE CHB - First Investigation in Stopping Tenofovir Disoproxil Fumarate (TDF) Treatment After Long Term Virologic Suppression in HBeAg-negative Chronic Hepatitis B
Brief Title: Stopping TDF Treatment After Long Term Virologic Suppression in HBeAg-negative CHB
Acronym: FINITE CHB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-EU-174-0160; 2010-021925-12 (EudraCT Number)
Record Dates: First submitted 2011-03-09; First posted 2011-03-23 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis B
Keywords: stopping oral antiviral therapy; HBsAg loss; seroconversion; restarting oral antiviral therapy
MeSH Terms: conditions — Hepatitis B, Chronic; HIV Seropositivity | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stop TDF (Experimental): Participants randomized to this arm will stop TDF therapy at baseline.
  Interventions: Other: Stop TDF
- Continue TDF (Active Comparator): Participants randomized to this arm will continue TDF therapy.
  Interventions: Drug: TDF

INTERVENTIONS:
Drug: TDF — Tenofovir disoproxil fumarate (TDF) 300 mg tablet administered orally once daily
  Other Names: Viread®
  Arms: Continue TDF
Other: Stop TDF — Participants will stop TDF therapy
  Arms: Stop TDF

SUMMARY:
The primary objective of this study is to evaluate hepatitis B surface antigen (HBsAg) loss and seroconversion in participants who stop tenofovir disoproxil fumarate (TDF) (Stop TDF arm) compared to participants who continue TDF (Continue TDF arm).

Only participants who already are on treatment with TDF monotherapy or TDF in combination with lamivudine or emtricitabine for at least 4 years and who achieved and maintained virologic suppression (< 400 copies/mL) for 3.5 or more years will be included in this study. One treatment arm will stop the TDF therapy while the other treatment arm will continue the TDF therapy. Participants in the Stop TDF arm will be monitored very closely with special focus on biochemical flares (especially alanine aminotransferase (ALT) increases) and virological relapses (Hepatitis B viral load increases). If any participant in the Stop TDF arm exceeds one or more predefined limits for such flares or relapses, TDF treatment will be reinstituted.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic hepatitis B, hepatitis B e-antigen negative, hepatitis B e-antibody positive, and hepatitis B surface antigen-positive
* Hepatitis B e Antigen (HBeAg)-negative at the beginning of TDF therapy (i.e. TDF monotherapy or combination of TDF + lamivudine or TDF + emtricitabine)
* Received continuous TDF therapy (i.e. TDF monotherapy or combination of TDF + lamivudine or TDF + emtricitabine) treatment for at least 4 years prior to screening. If TDF has been used in combination with lamivudine or emtricitabine, lamivudine or emtricitabine must have been stopped at least 12 weeks prior to screening
* Documented hepatitis B virus DNA (HBV DNA) < 400 copies/mL for at least 3.5 years prior to screening and at screening
* ALT within normal range
* α-fetoprotein (AFP) <= 50 ng/mL
* Calculated creatinine clearance >= 70 mL/min by Cockcroft-Gault formula using ideal body weight
* <= 10 kPa on Fibroscan assessment
* A negative serum pregnancy test for female subjects
* Adult subjects >= 18 years of age

Key Exclusion Criteria:

* Known cirrhosis
* Evidence of fibrosis >= Stage 3 (METAVIR) on liver biopsy or Fibroscan > 10 kPa within 6 months prior to screening
* Documentation of confirmed episodes (i.e., 2 consecutive values) of HBV DNA > 400 copies/mL within 3.5 years prior to screening
* History of decompensated liver disease (defined as direct [conjugated] bilirubin > 1.5 x upper limit of normal, prothrombin time (PT) > 1.5 x upper limit of normal, platelets < 75,000/mm³, serum albumin < 3.0 g/dL
* History of clinical hepatic decompensation in the judgement of the investigator
* Evidence of hepatocellular carcinoma
* Significant bone disease (in the judgment of the investigator)
* Serological evidence of coinfection with human immunodeficiency virus (HIV), hepatitis C virus, or hepatitis D infection
* Known hypersensitivity to TDF, its metabolites, or formulation excipients
* Concomitant therapy with disallowed medications
* History of malignant disease
* Lactating females
* Females wishing to became pregnant during the duration of the stud
* Subjects participating in another clinical trial can only be enrolled at the discretion of the Medical Monitor

Note: Other protocol defined inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-04-26 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- Germany (13):
  - Leberzentrum am Checkpoint, Berlin
  - Charite CVK, Berlin
  - Zentrum für HIV und Hepatitis, Düsseldorf
  - J.W. Goethe Universitaetsklinikum, Frankfurt
  - ifi Studien und Projekte GmbH, Hamburg
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinik Heidelberg, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis, Herne
  - Universitaetsklinikum Leipzig, Leipzig
  - Gemeinschaftspraxis Gastroenterologie, Leverkusen
  - Klinikum der LMU Grosshadern, München
  - Universitaetsklinikum Ulm, Ulm

REFERENCES:
- [Result] Berg T, Schott E, Felten G, Eisenbach C, Welzel TM, Warger T, et al. Stopping TDF Treatment After Long Term Virologic Suppression in HBeAg-Negative CHB: Two Cases From an Ongoing Randomized, Controlled Trial [Poster Number P47] The Viral Hepatitis Congress; 2012 September 7-9; Frankfurt am Main, Germany.
- [Result] Berg T, Simon K-G, Mauss S, Schott E, Heyne R, Klass D, et al. Stopping Tenofovir Disoproxil Fumarate Treatment After Long-Term Virologic Suppression in HBeAg-Negative CHB: Week 48 Interim Results From an Ongoing Randomized, Controlled Trial ("FINITE CHB") [Presentation P119]. The European Association for the Study of the Liver (EASL). 50th International Liver Congress; 2015 22-26 April; Vienna, Austria.
- [Derived] Berg T, Simon KG, Mauss S, Schott E, Heyne R, Klass DM, Eisenbach C, Welzel TM, Zachoval R, Felten G, Schulze-Zur-Wiesch J, Cornberg M, Op den Brouw ML, Jump B, Reiser H, Gallo L, Warger T, Petersen J; FINITE CHB study investigators [First investigation in stopping TDF treatment after long-term virological suppression in HBeAg-negative chronic hepatitis B]. Long-term response after stopping tenofovir disoproxil fumarate in non-cirrhotic HBeAg-negative patients - FINITE study. J Hepatol. 2017 Nov;67(5):918-924. doi: 10.1016/j.jhep.2017.07.012. Epub 2017 Jul 21. PMID 28736139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 13 study sites in Germany. The first participant was screened on 26 April 2011. The last study visit occurred on 23 August 2016.
Pre-assignment Details: 65 participants were screened.
Groups:
- Stop TDF: Participants stopped tenofovir disoproxil fumarate (Viread®; TDF) monotherapy at baseline.
- Continue TDF: Participants continued TDF monotherapy 300 mg once daily.
Period: Overall Study
Arm/Group | Stop TDF | Continue TDF
Started | 21 (13 participants did not restart TDF; 8 participants restarted TDF during the study.) | 22
Completed | 20 | 20
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Randomized but not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were either randomized to Arm A (Stop TDF) and had a baseline visit, or who were randomized to Arm B (Continue TDF) and received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Stop TDF | Continue TDF | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.51) | 45.0 (7.06) | 44.8 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 18 | 15 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 1 | 0 | 1
  White | 18 | 19 | 37
  Other | 1 | 1 | 2
Hepatitis B Virus Surface Antigen [Mean (Standard Deviation); unit: log10 IU/mL] | 4.4 (0.71) | 4.5 (0.35) | 4.5 (0.56)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With HBsAg Loss at Week 144 in Both Study Arms
Description: HBsAg loss is defined as qualitative HBsAg result changing from positive at baseline (BL) to negative at any post-baseline visit. Proportions are based on a Kaplan-Meier estimate.
Time Frame: Week 144
Population: HBsAg Loss and Seroconversion Full Analysis Set: participants in the Full Analysis Set who had at least one post-baseline HBsAg value and with HBsAg positive and HBsAb negative or missing at baseline.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Stop TDF: Participants stopped tenofovir disoproxil fumarate monotherapy at baseline.
Arm/Group | Stop TDF | Continue TDF
Number analyzed (Participants) | 21 | 21
Proportion of participants | 0.236 [0.095 to 0.516] | 0 [NA to NA] — No participants in the Continue TDF group had HBsAg loss.
Statistical Analysis 1: Comparison: Stop TDF vs Continue TDF; Test type: Superiority; p = 0.022, Log Rank — Log-rank test statistic was used to compare the time to HBsAg loss between the two treatment arms

2. Secondary Outcome: Proportion of Participants With HBsAg Seroconversion in Both Study Arms at Weeks 96 and 144
Description: HBsAg seroconversion is defined as qualitative HBsAb result changing from negative at baseline to positive at any postbaseline visit. Proportions are based on the Kaplan-Meier estimate.
Time Frame: Weeks 96 and 144
Population: HBsAg Loss and Seroconversion Full Analysis Set: participants in the Full Analysis Set who had at least 1 post-baseline HBsAg value and with HBsAg positive and HBsAb negative or missing at baseline.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Stop TDF | Continue TDF
Number analyzed (Participants) | 21 | 21
Proportion of participants
  HBsAg Seroconversion at Week 96 | 0.056 [0.008 to 0.334] | 0 [NA to NA] — No participants in the Continue TDF arm achieved HBsAg seroconversion at Week 96
  HBsAg Seroconversion at Week 144 | 0.203 [0.069 to 0.513] | 0 [NA to NA] — No participants in the Continue TDF arm achieved HBsAg seroconversion at Week 144

3. Secondary Outcome: Change From Baseline in Quantitative HBsAg (IU/mL) in Both Study Arms
Description: * The analyses were summarized by 3 treatment subgroups: Stop TDF (TDF-Free), Restart TDF, and Continue TDF
  * When participant randomized in the Stop TDF group restarted TDF therapy, that participant was considered part of the Restart TDF group from that point forward. For Restart TDF group, baseline is defined as the last available record on or prior to the restart date of TDF.
Time Frame: Baseline to Week 144
Population: Participants in the Full Analysis Set ( participants who were randomized to Stop TDF arm and had a baseline visit or who were randomized to Continue TDF arm and received at least 1 dose of study drug) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Stop TDF (TDF-Free): Participants who stopped TDF monotherapy at baseline. Participants in this group were TDF free.
- Restart TDF: Stop TDF participants who restarted TDF therapy
- Continue TDF: Participants who continued TDF monotherapy 300 mg once daily.
Arm/Group | Stop TDF (TDF-Free) | Restart TDF | Continue TDF
Number analyzed (Participants) | 21 | 8 | 21
log10 IU/mL
  Change from Baseline at Week 2: number analyzed (Participants) | 21 | 0 | 21
  Change from Baseline at Week 2 | -0.03 (0.139) |  | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 2.
  Change from Baseline at Week 4: number analyzed (Participants) | 20 | 0 | 20
  Change from Baseline at Week 4 | -0.03 (0.170) |  | -0.01 (0.105)
  Change from Baseline at Week 6: number analyzed (Participants) | 20 | 0 | 21
  Change from Baseline at Week 6 | -0.02 (0.192) |  | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 6.
  Change from Baseline at Week 8: number analyzed (Participants) | 20 | 0 | 21
  Change from Baseline at Week 8 | 0.04 (0.500) |  | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 8.
  Change from Baseline at Week 10: number analyzed (Participants) | 20 | 0 | 21
  Change from Baseline at Week 10 | 0.01 (0.556) |  | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 10.
  Change from Baseline at Week 12: number analyzed (Participants) | 19 | 1 | 21
  Change from Baseline at Week 12 | -0.11 (0.621) | -0.03 | -0.02 (0.137)
  Change from Baseline at Week 16: number analyzed (Participants) | 19 | 2 | 21
  Change from Baseline at Week 16 | -0.35 (0.741) | -0.73 (0.438) | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 16.
  Change from Baseline at Week 20: number analyzed (Participants) | 18 | 1 | 21
  Change from Baseline at Week 20 | -0.48 (0.949) | -0.42 | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 20.
  Change from Baseline at Week 24: number analyzed (Participants) | 18 | 2 | 21
  Change from Baseline at Week 24 | -0.56 (1.029) | -1.41 (1.211) | -0.07 (0.139)
  Change from Baseline at Week 28: number analyzed (Participants) | 17 | 3 | 21
  Change from Baseline at Week 28 | -0.60 (0.969) | -0.88 (0.916) | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 28.
  Change from Baseline at Week 32: number analyzed (Participants) | 16 | 3 | 21
  Change from Baseline at Week 32 | -0.77 (1.126) | -0.96 (1.211) | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 32.
  Change from Baseline at Week 36: number analyzed (Participants) | 17 | 2 | 21
  Change from Baseline at Week 36 | -0.67 (1.151) | -0.26 (0.461) | -0.08 (0.140)
  Change from Baseline at Week 40: number analyzed (Participants) | 18 | 3 | 21
  Change from Baseline at Week 40 | -0.78 (1.198) | -0.97 (1.275) | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 40.
  Change from Baseline at Week 44: number analyzed (Participants) | 17 | 1 | 21
  Change from Baseline at Week 44 | -0.87 (1.238) | -0.59 | NA (NA) — HBsAg assessment in the Continue TDF arm was not performed at Week 44.
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 3 | 20
  Change from Baseline at Week 48 | -0.88 (1.314) | -1.01 (1.295) | -0.11 (0.101)
  Change from Baseline at Week 60: number analyzed (Participants) | 18 | 3 | 21
  Change from Baseline at Week 60 | -0.96 (1.353) | -1.03 (1.236) | -0.10 (0.133)
  Change from Baseline at Week 72: number analyzed (Participants) | 16 | 5 | 20
  Change from Baseline at Week 72 | -1.22 (1.478) | -0.64 (1.085) | -0.14 (0.142)
  Change from Baseline at Week 84: number analyzed (Participants) | 16 | 5 | 21
  Change from Baseline at Week 84 | -1.21 (1.555) | -0.69 (1.084) | -0.16 (0.164)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 5 | 20
  Change from Baseline at Week 96 | -1.22 (1.530) | -0.69 (1.031) | -0.17 (0.159)
  Change from Baseline at Week 108: number analyzed (Participants) | 16 | 5 | 20
  Change from Baseline at Week 108 | -1.43 (1.573) | -0.69 (1.088) | -0.17 (0.145)
  Change from Baseline at Week 120: number analyzed (Participants) | 14 | 7 | 20
  Change from Baseline at Week 120 | -1.56 (1.752) | -0.58 (0.870) | -0.20 (0.136)
  Change from Baseline at Week 132: number analyzed (Participants) | 13 | 7 | 20
  Change from Baseline at Week 132 | -1.74 (1.829) | -0.52 (0.941) | -0.22 (0.172)
  Change from Baseline at Week 144: number analyzed (Participants) | 13 | 8 | 20
  Change from Baseline at Week 144 | -1.80 (1.796) | -0.51 (0.861) | -0.22 (0.160)

4. Secondary Outcome: Proportion of Participants Who Restart TDF Therapy in the Stop TDF Arm
Time Frame: Weeks 48, 96, and 144
Population: Full Analysis Set (FAS): participants who were randomized to Stop TDF group and had a baseline visit or who were randomized to Continue TDF group and received at least 1 dose of study drug. Proportions are based on the Kaplan-Meier estimate.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Stop TDF: Participants stopped TDF monotherapy at baseline.
Arm/Group | Stop TDF
Number analyzed (Participants) | 21
Proportion of participants
  TDF Restart at Week 48 | 0.143 [0.048 to 0.380]
  TDF Restart at Week 96 | 0.238 [0.107 to 0.481]
  TDF Restart at Week 144 | 0.381 [0.212 to 0.619]

5. Secondary Outcome: Percentage of Participants With Viral Suppression in the Stop TDF Arm (TDF-Free and Re-Start TDF Groups)
Description: Viral suppression is defined as 2 consecutive assessments of HBV DNA < 400 copies/mL (69 IU/mL) through Week 144.
Time Frame: Baseline to Week 144
Population: Participants in the FAS with available data were analyzed. When participant randomized in the Stop TDF group restarted TDF therapy, that participant was considered part of the Restart TDF group from that point forward. 1 participant restarted TDF during Wk 72, thus was reported in both Stop TDF and Restart TDF arms based on the TDF restart date.
Measure: Number; unit: Percentage of participants
Groups:
- Stop TDF (TDF-Free): Participants stopped TDF monotherapy at baseline. Participants in this group were TDF free.
- Re-Start TDF: Stop TDF participants who restarted TDF therapy
Arm/Group | Stop TDF (TDF-Free) | Re-Start TDF
Number analyzed (Participants) | 21 | 8
Percentage of participants
  Week 2: number analyzed (Participants) | 21 | 0
  Week 2 | 52.4 |
  Week 4: number analyzed (Participants) | 19 | 0
  Week 4 | 5.3 |
  Week 6: number analyzed (Participants) | 20 | 0
  Week 6 | 10.0 |
  Week 8: number analyzed (Participants) | 20 | 0
  Week 8 | 5.0 |
  Week 10: number analyzed (Participants) | 20 | 0
  Week 10 | 15.0 |
  Week12: number analyzed (Participants) | 19 | 1
  Week12 | 21.1 | 0
  Week 16: number analyzed (Participants) | 19 | 2
  Week 16 | 31.6 | 0
  Week 20: number analyzed (Participants) | 18 | 2
  Week 20 | 27.8 | 0
  Week 24: number analyzed (Participants) | 18 | 2
  Week 24 | 16.7 | 0
  Week 28: number analyzed (Participants) | 17 | 3
  Week 28 | 17.6 | 0
  Week 32: number analyzed (Participants) | 16 | 3
  Week 32 | 12.5 | 66.7
  Week 36: number analyzed (Participants) | 17 | 2
  Week 36 | 29.4 | 100.0
  Week 40: number analyzed (Participants) | 18 | 3
  Week 40 | 22.2 | 100.0
  Week 44: number analyzed (Participants) | 17 | 1
  Week 44 | 29.4 | 100.0
  Week 48: number analyzed (Participants) | 18 | 3
  Week 48 | 27.8 | 100.0
  Week 60: number analyzed (Participants) | 18 | 3
  Week 60 | 33.3 | 100.0
  Week 72: number analyzed (Participants) | 17 | 5
  Week 72 | 35.3 | 60.0
  Week 84: number analyzed (Participants) | 16 | 5
  Week 84 | 31.3 | 100.0
  Week 96: number analyzed (Participants) | 16 | 5
  Week 96 | 37.5 | 100.0
  Week 108: number analyzed (Participants) | 16 | 5
  Week 108 | 37.5 | 100.0
  Week 120: number analyzed (Participants) | 15 | 7
  Week 120 | 40.0 | 71.4
  Week 132: number analyzed (Participants) | 13 | 7
  Week 132 | 38.5 | 100.0
  Week 144: number analyzed (Participants) | 13 | 8
  Week 144 | 46.2 | 87.5

6. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) > Upper Limit of the Normal Range in the Stop TDF Arm (TDF-Free and Restart TDF)
Time Frame: Baseline to Week 144
Population: Participants in the Full Analysis Set with available data were analyzed. Percentages are based on the number of participants with non-missing laboratory test results at each visit. One participant restarted TDF during Weeks 72 and 120 and thus was reported in both the Stop TDF and Re-Start TDF groups based on the date of TDF restart.
Measure: Number; unit: Percentage of participants
Arm/Group | Stop TDF (TDF-Free) | Re-Start TDF
Number analyzed (Participants) | 21 | 8
Percentage of participants
  Week 2: number analyzed (Participants) | 21 | 0
  Week 2 | 4.8 |
  Week 4: number analyzed (Participants) | 20 | 0
  Week 4 | 0 |
  Week 6: number analyzed (Participants) | 20 | 0
  Week 6 | 35.0 |
  Week 8: number analyzed (Participants) | 20 | 0
  Week 8 | 60.0 |
  Week 10: number analyzed (Participants) | 20 | 0
  Week 10 | 70.0 |
  Week 12: number analyzed (Participants) | 19 | 2
  Week 12 | 42.1 | 100.0
  Week 16: number analyzed (Participants) | 19 | 2
  Week 16 | 26.3 | 100.0
  Week 20: number analyzed (Participants) | 17 | 2
  Week 20 | 11.8 | 100.0
  Week 24: number analyzed (Participants) | 18 | 2
  Week 24 | 16.7 | 50.0
  Week 28: number analyzed (Participants) | 17 | 3
  Week 28 | 11.8 | 33.3
  Week 32: number analyzed (Participants) | 15 | 3
  Week 32 | 13.3 | 0
  Week 36: number analyzed (Participants) | 17 | 2
  Week 36 | 11.8 | 0
  Week 40: number analyzed (Participants) | 17 | 3
  Week 40 | 23.5 | 0
  Week 44: number analyzed (Participants) | 17 | 1
  Week 44 | 11.8 | 0
  Week 48: number analyzed (Participants) | 18 | 3
  Week 48 | 16.7 | 0
  Week 60: number analyzed (Participants) | 18 | 3
  Week 60 | 22.2 | 0
  Week 72: number analyzed (Participants) | 17 | 5
  Week 72 | 11.8 | 40
  Week 84: number analyzed (Participants) | 16 | 5
  Week 84 | 18.8 | 0
  Week 96: number analyzed (Participants) | 16 | 5
  Week 96 | 12.5 | 0
  Week 108: number analyzed (Participants) | 16 | 5
  Week 108 | 18.8 | 0
  Week 120: number analyzed (Participants) | 15 | 7
  Week 120 | 20.0 | 14.3
  Week 132: number analyzed (Participants) | 12 | 7
  Week 132 | 0 | 28.6
  Week 144: number analyzed (Participants) | 13 | 8
  Week 144 | 15.4 | 0

7. Secondary Outcome: Proportion of Participants With HBsAg Loss at Week 96 in Both Study Arms
Description: as for outcome 1
Time Frame: Week 96
Population: HBsAg Loss and Seroconversion Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Stop TDF | Continue TDF
Number analyzed (Participants) | 21 | 21
Proportion of participants | 0.172 [0.058 to 0.446] | 0 [NA to NA] — No participants in the Continue TDF group had HBsAg loss

ADVERSE EVENTS:
Time Frame: Up to 144 weeks
Description: * Safety Analysis Set
  * TDF-emergent Events (Restart TDF and Continue TDF): events began on/after date of TDF restart until last dose day for subjects who restarted TDF in the Stop TDF group and on/after Study Day 1 until last dose day for subjects in the Continue TDF group
  * Termination-emergent Events (TDF-Free): events began on/after Study Day 1 for the Stop TDF group until last study day for subjects who did not restart TDF and prior to date of restart for subjects who restarted TDF
Groups:
- Stop TDF (TDF-Free) [Termination Emergent]: Participants stopped TDF monotherapy at baseline.
- Re-start TDF [TDF Emergent]: Stop TDF participants who restarted TDF therapy.
- Continue TDF [TDF Emergent]: Participants continued TDF monotherapy 300 mg once daily.
Arm/Group | Stop TDF (TDF-Free) [Termination Emergent] | Re-start TDF [TDF Emergent] | Continue TDF [TDF Emergent]
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/8 | 0/21
Serious Adverse Events (participants affected / at risk) | 4/21 | 1/8 | 3/21
Other Adverse Events (participants affected / at risk) | 17/21 | 6/8 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stop TDF (TDF-Free) [Termination Emergent] (N=21) | Re-start TDF [TDF Emergent] (N=8) | Continue TDF [TDF Emergent] (N=21)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Surgical failure (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stop TDF (TDF-Free) [Termination Emergent] (N=21) | Re-start TDF [TDF Emergent] (N=8) | Continue TDF [TDF Emergent] (N=21)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 2
Influenza like illness (General disorders) | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 11 | 1 | 6
Sinusitis (Infections and infestations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Headache (Nervous system disorders) | 5 | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years